CLINICAL TRIAL: NCT02844244
Title: Training Workshop for Promoting Family Health, Happiness and Harmony Through a Community-based "Learning Families" Campaign
Brief Title: Training Workshop for Promoting Family Well-being Through a Community-based "Learning Families" Campaign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Christian Family Service Centre (Other); The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UW10-415
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Family; Well-being
Keywords: family well-being; positive psychology
MeSH Terms: interventions — Sensitivity Training Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- training group (Experimental): Two two-hour training sessions for the participants. It aimed to train lay resident leaders to be peer health promoters. The peer health promoters were taught either to independently implement or to assist social workers to conduct a series of community-based family well-being activities.
  Interventions: Behavioral: training group

INTERVENTIONS:
Behavioral: training group — The training workshop included two two-hour sessions. It focused on the enhancement of knowledge, attitude, and practice of peer health promoters on implementing community activities for the residents.

SUMMARY:
To strengthen family well-being and neighborhood cohesion in Kwun Tong community, a community -based "Learning families" campaign was conducted. As an initial step of this project, the investigators conducted a need assessments before designing and conducting a train-the-trainer workshop.The train-the-trainer workshop aimed to prepare the members of Estate Management Advisory Committees (EMAC) and Mutual Aid Committees (MACs) to implement and assist in conducting a series of community-based family well-being activities for residents in a public housing estate. Focus group interviews (before and one year after training workshop) were conducted to obtain opinion from the members of EMAC and MACs of the public housing estate. Questionnaire assessments were conducted before, immediately after finishing the training workshop, one year after training workshop.

DETAILED DESCRIPTION:
According to the Social Welfare Department statistics, Kwun Tong has been ranked as the highest for the reported cases of elderly abuse (12.3%), the second and fourth highest for the reported cases of battered spouse (9.2%) and child abuse (7.9%) respectively . To strengthen family well-being in the Kwun Tong community, the investigators adopt a community-based participatory (CBP) approach and implement a community-based "Learning Families" campaign in Kwun Tong district with our collaborator, the Christian Family Service Centre (CFSC). The campaign aims to promote family health, happiness, and harmony (3Hs) through cultivating cooperative and self-regulated family learning culture in the public housing estate

Given that CFSC is the leading non-government organization based in Kwun Tong district, the investigators believe that the proposed campaign will deliver the family well-being messages effectively in the community via engaging major stakeholders such as the Estate Management Advisory Committees (EMACs) and the Mutual Aid Committees (MACs).

The investigators implemented a brief training sessions to the resident leaders of EMAC & MACs to engage and equip them with the general concept of "Family well-being", " Learning family", "Neighbourhood cohesion" and activities organizing skills. The train-the-trainer workshop aimed to prepare the members of Estate Management Advisory Committees (EMAC) and Mutual Aid Committees (MACs) to implement and assist in conducting a series of community-based family well-being activities for residents in a public housing estate.

Focus group interviews (before and one year after training workshop) were conducted to obtain opinion from the members of EMAC and MACs of the public housing estate. Questionnaire assessments were conducted before, immediately after finishing the training workshop, one year after training workshop.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese older 18 years of age,
* able to read Chinese and speak Cantonese,
* willing to carry out the duties of peer health promoters in the project.

Exclusion Criteria:

- not fit the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in learning | Baseline, immediately after finishing training workshop "up to 30 min" and one year after training workshop
  Assessed by outcome-based questionnaire

SECONDARY OUTCOMES:
Reactions to training content | Immediately after finishing training workshop "up to 30 min" and one year after training workshop
  Assessed by outcome-based questionnaire
Practice of implementing community activities | Baseline and one year after training workshop
  Assessed by outcome-based questionnaire
change the residents' family well-being | Baseline and one year after training workshop
  Assessed by outcome-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Study Director — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Layne JE, Sampson SE, Mallio CJ, Hibberd PL, Griffith JL, Das SK, Flanagan WJ, Castaneda-Sceppa C. Successful dissemination of a community-based strength training program for older adults by peer and professional leaders: the people exercising program. J Am Geriatr Soc. 2008 Dec;56(12):2323-9. doi: 10.1111/j.1532-5415.2008.02010.x. PMID 19112654
- [Background] McClelland JW, Irving LM, Mitchell RE, Bearon LB, Webber KH. Extending the reach of nutrition education for older adults: feasibility of a Train-the-Trainer approach in congregate nutrition sites. J Nutr Educ Behav. 2002 Mar-Apr;34 Suppl 1:S48-52. doi: 10.1016/s1499-4046(06)60311-4. PMID 12047829
- [Background] Forst L, Lacey S, Chen HY, Jimenez R, Bauer S, Skinner S, Alvarado R, Nickels L, Zanoni J, Petrea R, Conroy L. Effectiveness of community health workers for promoting use of safety eyewear by Latino farm workers. Am J Ind Med. 2004 Dec;46(6):607-13. doi: 10.1002/ajim.20103. PMID 15551366
- [Background] Sin NL, Lyubomirsky S. Enhancing well-being and alleviating depressive symptoms with positive psychology interventions: a practice-friendly meta-analysis. J Clin Psychol. 2009 May;65(5):467-87. doi: 10.1002/jclp.20593. PMID 19301241
- [Derived] Lai AY, Stewart SM, Wan A, Fok H, Lai HYW, Lam TH, Chan SS. Development and evaluation of a training workshop for lay health promoters to implement a community-based intervention program in a public low rent housing estate: The Learning Families Project in Hong Kong. PLoS One. 2017 Aug 25;12(8):e0183636. doi: 10.1371/journal.pone.0183636. eCollection 2017. PMID 28841677